CLINICAL TRIAL: NCT06155565
Title: Investigating Patterns in Enrollment and Engagement Among Individuals Coping With Anxiety Disorder
Brief Title: Understanding Patient Engagement Trends in Anxiety Disorder Clinical Research
Status: Not yet recruiting | Type: Observational
Sponsor: Power Life Sciences Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 65829005
Record Dates: First submitted 2023-11-24; First posted 2023-12-04 (Actual); Last update posted 2023-12-04 (Actual); Status verified 2023-11

CONDITIONS: Anxiety Disorder
Keywords: anxiety disorder
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Clinical trials, specifically focused on anxiety disorder, are crucial in assessing the safety and efficacy of new treatments. These trials serve as fundamental instruments in determining whether emerging medications outperform standard therapies, providing compelling evidence to support wider implementation.

The main goal is to thoroughly scrutinize trial completion rates and voluntary withdrawals among this particular group of patients.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 18 years old
* Diagnosis of anxiety disorder
* Able to comprehend the investigational nature of the protocol and provide informed consent

Exclusion Criteria:

* Female patients who are currently pregnant or nursing
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Inability to perform regular electronic reporting

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with anxiety disorder who are actively considering enrolling in a clinical study for said condition, but have not yet completed enrollment and randomization.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-12 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Number of anxiety disorder patients who decide to enroll in a clinical research | 3 months
Rate of anxiety disorder patients who remain in clinical trial to trial completion | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Gill, Study Director — Power Life Sciences Inc.
Locations (1):
- Power Life Sciences, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Szuhany KL, Simon NM. Anxiety Disorders: A Review. JAMA. 2022 Dec 27;328(24):2431-2445. doi: 10.1001/jama.2022.22744. PMID 36573969
- [Background] Yee A, Ng CG, Seng LH. Vortioxetine Treatment for Anxiety Disorder: A Meta-Analysis Study. Curr Drug Targets. 2018;19(12):1412-1423. doi: 10.2174/1389450118666171117131151. PMID 29149828
- [Background] Liao J, Kang J, Li F, Li Q, Wang J, Tang Q, Mao N, Li S, Xie X. A cross-sectional study on the association of anxiety and depression with the disease activity of systemic lupus erythematosus. BMC Psychiatry. 2022 Sep 5;22(1):591. doi: 10.1186/s12888-022-04236-z. PMID 36064377

DOCUMENTS (1):
  • Informed Consent Form (2023-11-24): https://cdn.clinicaltrials.gov/large-docs/65/NCT06155565/ICF_000.pdf